CLINICAL TRIAL: NCT01880047
Title: Safety and Efficacy of Eltrombopag at Escalated Doses up to 150mg in Patients With Persistent and Chronic Immune Thrombocytopenia (ITP) Not Responsive to 75 mg
Brief Title: Safety and Efficacy of Eltrombopag at Escalated Doses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116862
Record Dates: First submitted 2012-11-20; First posted 2013-06-18 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Immune Thrombocytopenia; Platelet Disorder
Keywords: Immune Thrombocytopenia; ITP; Eltrombopag; Promacta
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Blood Platelet Disorders | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eltrombopag (Active Comparator): Subjects in the study will receive 75 mg eltrombopag and then be randomized to receive either an additional 25 mg of eltrombopag or matching placebo tablet dispensed by the research pharmacy. Subjects and investigators will be blinded to randomization. Randomization will be stratified according to splenectomy status. Randomization will be performed at the time of informed consent with a computer generated randomization table. Subjects and investigators will be blinded to assignment and treatment in this phase.
  Interventions: Drug: Eltrombopag
- Placebo (Placebo Comparator): Subjects will be randomly allocated in a two to one ratio to receive treatment or placebo. All subjects in the study will receive 75 mg eltrombopag and then be randomized to receive either an additional 25 mg of eltrombopag or matching placebo tablet dispensed by the research pharmacy. Subjects and investigators will be blinded to randomization. Randomization will be stratified according to splenectomy status.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag will be administered for 8 weeks or until the platelet count exceeds 150,000; at this point dosing will stop, subject will be considered a responder and the subject will eligible for entering Part 2 (the long term treatment part of the study. The dose at which the subject achieved the primary endpoint (> 50,000 and increase by > 20,000) will be considered the dose of response. Dose escalation will continue, despite satisfaction of the primary endpoint of study (> 50,000 and > 20,000 above baseline), unless the platelet count reaches the lower limit of normal range 150,000. Subjects will stop study medication if the platelet count is within the normal range, thereby minimizing any safety risk associated with elevated platelet count.
  Other Names: SB-497115-GR; Promacta
  Arms: Eltrombopag
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study rationale is based on the data that in previous clinical studies of eltrombopag in ITP there are some patients who have been reported as non responders at the maximal approved dose of 75 mg daily. The trend in both normal volunteers and in patients with ITP suggest and increasing response rate with increased doses of eltrombopag up to a dose of 75mg. Previously published data has shown no overt increase in toxicity in normal volunteers, oncology patients and aplastic anemia patients treated with escalated doses as high or higher than those proposed in this study.

It therefore seems possible that in ITP patients who did not respond to a dose of 75mg daily, eltrombopag could be more effective at a higher dose. We propose a double blind randomized controlled trial in ITP patients who have been defined as non-responders at the maximum dose (75mg) of eltrombopag, assessing efficacy and toxicity at higher daily doses (100mg, 125 mg, 150 mg)

DETAILED DESCRIPTION:
Preliminary data in pediatric patients (who seem to metabolize eltrombopag differently especially at younger ages) find that in the middle and lowest age cohort, even doses of 75 mg were often insufficient to obtain a response.

Altogether, this data suggest both that a higher dose in ITP may be more efficacious in increasing the platelet count and that there is no overt increase in toxicity in normal volunteers, oncology patients and aplastic anemia patients treated with doses as high or higher than those proposed in this study.

Double-blind, randomized, placebo-controlled trial in subjects with ITP who are 'non-responders' at the maximum package insert dose (75mg) of eltrombopag; non-responders are those with platelet counts < 50,000 despite taking 75 mg/day of eltrombopag for at least 3 weeks.

Study Design (First part): 8 Weeks

Subjects will be randomly allocated in a two to one ratio to receive treatment or placebo. All subjects in the study will receive 75 mg eltrombopag and then be randomized to receive either an additional 25 mg of eltrombopag or matching placebo tablet dispensed by the research pharmacy. Subjects and investigators will be blinded to randomization. Randomization will be stratified according to splenectomy status. Randomization will be performed at the time of informed consent with a computer generated randomization table. Subjects and investigators will be blinded to assignment and treatment in this phase. Eltrombopag will be administered for 8 weeks or until the platelet count exceeds 100,000; at this point dosing will stop, subject will be considered a responder and the subject will eligible for entering Part 2 (the long term treatment part of the study) if desired and agreed to be appropriate by the subject giving consent, and the treating physician. The dose at which the subject achieved the primary endpoint (> 50,000 and increase by > 20,000) will be considered the dose of response. Even if a patient achieves a response, if the platelet counts remains < 100,000, then the dose escalation schema in the figure above will continue.

Dose escalation will continue, despite satisfaction of the primary endpoint of study (> 50,000 and > 20,000 above baseline), unless the platelet count reaches 100,000. The rationale for this approach is to maximize clinically relevant responses for the subjects and standardize data for analysis. Subjects will stop study medication if the platelet count is within the normal range, thereby minimizing any safety risk associated with elevated platelet count. By continuing to dose escalate subjects until the platelet count is > 100,000, the maximum response and correlation of dose will be tracked allowing better understanding of sustained response and dose-dependent response, which can be applied to future consideration dosage for periods of short-term hemostasis ( i.e surgical procedures). The 8 weeks of data collected in enrolled subjects on the standardized protocol will have the balance of consistency of dosage and unequivocality of response while maintaining subject safety.

Enrollment will be stratified to address concerns regarding the inclusion of pediatric subjects. Enrollment will begin with adult subjects ≥ 18 years of age, until there is safety information available for review from at least three adult patients who received active therapy for 8 weeks with exposure to the maximal proposed dose of 150 mg. After review of this unblinded safety information by independent Data Safety Monitoring Officer (DMSO) we will allow pediatric patients 12-18 years of age to enroll on the protocol.

Long Term Treatment Extension (Part 2): (18 months)

After 8 weeks or once dosing is stopped because the platelet count is > 100,000, the subject will be unblinded, once the data forms are complete with the assistance of the research pharmacy.

Subjects who received and responded to eltrombopag higher dose treatment will have the option to continue therapy with periodic monitoring and ongoing dose adjustment.

Subject who had a platelet count > 100,000 can enter Part 2 at the dose at which the subject met primary response criteria after the platelet count decreases to < 100,000/uL (microliters) on serial monitoring in the immediate post-study monitoring period.

Subjects randomized to the placebo group who did not respond will have the opportunity to receive open label escalated dose eltrombopag over 8 weeks following the study protocol as if they had been randomized to active drug in the study. This group will provide the "confirmatory group" to see if the rate of response in the randomized group can be confirmed in this group.

Consent will be obtained for additional monitoring with bone marrow aspirate and biopsy at 1 year and additional ophthalmologic examinations at 6 months and 18 months.

The trial will have an 80% statistical power at the 5% level of significance (two sided) to detect a difference in the proportion of subjects receiving increased dose of eltrombopag with a primary response (2 consecutive platelet counts of > 50,000 and an increase of > 20,000 from the study baseline with in the 8 week increased dose window not as a result of rescue treatment ) to subjects without a primary response in the placebo group assuming 50% of subjects randomized to active drug will have a response and 5% of subjects randomized to placebo would have a response. However an interim analysis would be performed after 18 subjects to test for futility and efficacy and also to re-estimate sample size. If neither futility or efficacy are met the trial would continue to enroll. Based on the observed treatment effect at the interim analysis the sample size would be allowed to expand to up to 60 subjects.

Dose modification will be made on the basis of individual platelet response as detailed below to a maximal dose of 150mg.

ELIGIBILITY:
Inclusion Criteria:

* Subject or their parent/ guardian has signed and dated a written informed consent
* Male and Females aged 12 years or older diagnosed with chronic ITP according to the new consensus guidelines
* No indication of a disease which may cause thrombocytopenia other than ITP----no specific testing required
* Subjects with thrombocytopenia ≤ 50,000 /uL after at least 21 days of daily dosage with eltrombopag 75mg
* Stable dosage of concomitant treatments for ITP

  ≥ 2 weeks or longer (corticosteroids);
* At least 2 weeks from rescue therapy for ITP (WinRho, Intravenous Immunoglobulin (IVIG), corticosteroids, platelet transfusion)
* At least 4 weeks from rituximab treatment
* Pregnant or Lactating Women are excluded
* Women of child-bearing age with a negative pregnancy test within 7 days of enrollment and who agree to use acceptable methods of birth control will be eligible for this study
* Female subjects or female partners of male subjects must either be of non-child bearing potential (hysterectomy, bilateral ovariectomy, bilateral tubal ligation or post menopausal for more than one year) OR, if of child bearing potential, using one of the following highly effective methods of contraception.
* complete abstinence from intercourse
* Intrauterine device (IUD)
* Two forms of barrier contraception. diaphragm plus spermicide, or for males condoms plus spermicide.
* Male partner is sterile and is the only partner of the female.
* Systemic contraceptives (combined oral progesterone only)

Exclusion Criteria:

* Previous history of eltrombopag-related liver function test (LFT) elevation that required interruption of treatment
* Previous history of immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to eltrombopag
* HIV Infection
* History of Arterial of Venous Thrombosis within the past year or requiring ongoing therapy
* Active Hepatitis C infection
* Treatment with medications that affect platelet function ( including but not limited to Aspirin, Clopidogrel and /or NSAIDs) or anti-coagulant medications
* Elevated Aspartate Aminotransferase(AST/ALT) or Creatinine > 1.5 times upper limit of normal in 4 weeks prior to enrollment*
* Abnormalities in white blood cell count (WBC), automatic neutrophil count (ANC), and Hemoglobin > 1.5 times upper or lower limit of normal*
* * Subjects can be rescreened to be included

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sujit Sheth, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One splenectomized subject was removed from the study because of increased bone marrow reticulin, prior to receiving any study drug
Groups:
- Non-Splenectomized Eltrombopag; Splenectomized Eltrombopag: Subjects randomized to this group were treated with 100 mg daily eltrombopag for 2 weeks, then escalated to 125 mg daily for 2 weeks and then to 150 mg daily for 4 weeks
- Non-Splenectomized Placebo; Splenectomized Placebo: Subjects randomized to this group were treated with 75 mg eltrombopag plus placebo for 8 weeks
Period: Weeks 0-2
Arm/Group | Non-Splenectomized Eltrombopag | Non-Splenectomized Placebo | Splenectomized Eltrombopag | Splenectomized Placebo
Started | 17 | 9 | 5 | 3
Completed | 17 | 8 | 4 | 2
Not Completed | 0 | 1 | 1 | 1
Period: Weeks 3-4
Arm/Group | Non-Splenectomized Eltrombopag | Non-Splenectomized Placebo | Splenectomized Eltrombopag | Splenectomized Placebo
Started | 17 | 8 | 4 | 2
Completed | 17 | 7 | 4 | 2
Not Completed | 0 | 1 | 0 | 0
Period: Weeks 5-8
Arm/Group | Non-Splenectomized Eltrombopag | Non-Splenectomized Placebo | Splenectomized Eltrombopag | Splenectomized Placebo
Started | 17 | 7 | 4 | 2
Completed | 15 | 6 | 4 | 2
Not Completed | 2 | 1 | 0 | 0
Period: Extension Phase - 18 Months
Arm/Group | Non-Splenectomized Eltrombopag | Non-Splenectomized Placebo | Splenectomized Eltrombopag | Splenectomized Placebo
Started | 15 (15 subjects went into extension phase, were followed for variable periods of time) | 6 (6 subjects went into extension phase, were followed for variable periods of time) | 4 (4 subjects went into extension phase, were followed for variable periods of time) | 2 (2 subjects went into extension phase, were followed for variable periods of time)
Completed | 6 | 3 | 3 | 0
Not Completed | 9 | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Subjects randomly assigned to the treatment or placebo arm in a 2:1 ratio as described
Groups:
- Non-splenectomized Active Drug: Includes patients on active drug who have not been splenectomized
- Non-splenectomized Placebo: Includes patients on placebo who have not been splenectomized
- Splectomized on Active Drug: Includes patients on active drug who have been splenectomized
- Splectomized on Placebo: Includes patients on placebo who have been splenectomized
- Total: Total of all reporting groups
Arm/Group | Non-splenectomized Active Drug | Non-splenectomized Placebo | Splectomized on Active Drug | Splectomized on Placebo | Total
Number analyzed (Participants) | 17 | 9 | 5 | 3 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 5 | 0 | 0 | 13
  Between 18 and 65 years | 8 | 1 | 3 | 3 | 15
  >=65 years | 1 | 3 | 2 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 3 | 3 | 18
  Male | 11 | 3 | 2 | 0 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 9 | 5 | 3 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Responding to >75mg Daily as Defined by a Rise in Platelet Count by 20,000/Microliter, With a Total Platelet Count >50,000/Microliter, ON TWO CONSECUTIVE OCCASIONS During the 8 Week Period
Description: To determine if patients with chronic ITP who do not respond to 75 mg of eltrombopag daily given for at least 3 weeks but then do respond to eltrombopag given daily first for 2 weeks at doses of 100, then for 2 weeks at 125 mg and finally for 4 weeks at a dose of 150mg daily. Response will be defined as 2 consecutive platelet counts of > 50,000 with an increase of > 20,000 from the study baseline within the 8 week increased dose window not as a result of rescue treatment.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Splenectomized Eltrombopag | Non-Splenectomized Placebo | Splenectomized Eltrombopag | Splenectomized Placebo
Number analyzed (Participants) | 15 | 6 | 4 | 2
Participants | 10 | 3 | 1 | 1

2. Secondary Outcome: Number of Particiapants With Drug Related Adverse Events
Description: Monitoring for AEs, SAEs, abnormalities in liver or kidney function, thrombotic complications, hematologic malignancies, parameters suggesting bone marrow fibrosis (a bone marrow may be done at the discretion of the investigator), cataracts.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Splenectomized Eltrombopag | Non-Splenectomized Placebo | Splenectomized Eltrombopag | Splenectomized Placebo
Number analyzed (Participants) | 15 | 6 | 4 | 2
Participants | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Data were collected over the 8 week primary study period
Description: Monitoring for AEs, SAEs, abnormalities in liver or kidney function, thrombotic complications, hematologic malignancies, parameters suggesting bone marrow fibrosis (a bone marrow may be done at the discretion of the investigator), cataracts.
Groups:
- Eltrombopag 100 mg: This group includes subjects on active drug (splenectomized and no-splenectomized who had adverse events at the 100 mg dose
- Eltombopag 125: This group includes subjects on active drug (splenectomized and no-splenectomized who had adverse events at the 125 mg dose
- Eltombopag 150: This group includes subjects on active drug (splenectomized and no-splenectomized who had adverse events at the 150 mg dose
- Placebo 100: This group includes subjects on placebo (splenectomized and no-splenectomized who had adverse events at the 100 mg dose
- Placebo 125: This group includes subjects on placebo (splenectomized and no-splenectomized who had adverse events at the 125 mg dose
- Placebo 150: This group includes subjects on placebo (splenectomized and no-splenectomized who had adverse events at the 150 mg dose
- Open Label Phase: Subjects included are those who were on placebo and those who were on eltrombopag, all at 150 mg dose
Arm/Group | Non-Splenectomized Eltrombopag | Non-Splenectomized Placebo | Splenectomized Eltrombopag | Splenectomized Placebo | Eltrombopag 100 mg | Eltombopag 125 | Eltombopag 150 | Placebo 100 | Placebo 125 | Placebo 150 | Open Label Phase
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/9 | 0/5 | 0/3 | 0/22 | 0/21 | 0/19 | 0/11 | 0/10 | 0/8 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/17 | 1/9 | 0/5 | 0/3 | 1/22 | 1/21 | 1/19 | 0/11 | 0/10 | 0/8 | 0/27
Other Adverse Events (participants affected / at risk) | 13/17 | 5/9 | 1/5 | 1/3 | 4/22 | 5/21 | 12/19 | 2/11 | 5/10 | 6/8 | 22/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Splenectomized Eltrombopag (N=17) | Non-Splenectomized Placebo (N=9) | Splenectomized Eltrombopag (N=5) | Splenectomized Placebo (N=3) | Eltrombopag 100 mg (N=22) | Eltombopag 125 (N=21) | Eltombopag 150 (N=19) | Placebo 100 (N=11) | Placebo 125 (N=10) | Placebo 150 (N=8) | Open Label Phase (N=27)
Increased liver enzymes >3 times ULN (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal Prolapse (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Splenectomized Eltrombopag (N=17) | Non-Splenectomized Placebo (N=9) | Splenectomized Eltrombopag (N=5) | Splenectomized Placebo (N=3) | Eltrombopag 100 mg (N=22) | Eltombopag 125 (N=21) | Eltombopag 150 (N=19) | Placebo 100 (N=11) | Placebo 125 (N=10) | Placebo 150 (N=8) | Open Label Phase (N=27)
Respiratory infection (Infections and infestations) | 10 (15) | 4 (7) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 4 (4) — Respiratory infection - Not related to study medication/placebo
Bleeding (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 1 (2) | 0 (0) | 3 (5) | 2 (3) | 6 (8) | 2 (4) | 3 (3) | 4 (6) | 16 (22) — Epistaxis
Transaminitis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (3) — Transaminitis not requiring study intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT01880047/Prot_SAP_000.pdf